CLINICAL TRIAL: NCT03209427
Title: Pruritus After Intrathecal Morphine in Cesarean Section: Incidence, Severity and Its Relation to Serum Serotonin Level
Brief Title: Serum Serotonin and Pruritus After Intrathecal Morphine in Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed galal aly, Assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17100209
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Pruritus
Keywords: morphine, pruritus, serotonin
MeSH Terms: conditions — Pruritus | interventions — Morphine; volociximab

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): intrathecal injection of 100 μg morphine
  Interventions: Drug: Morphine 100 μg
- Group II (Active Comparator): iIntrathecal injection of 200 μg morphine
  Interventions: Drug: Morphine 200 μg

INTERVENTIONS:
Drug: Morphine 100 μg — Intrathecal injection of morphine100 μg
  Other Names: M100
  Arms: Group I
Drug: Morphine 200 μg — Intrathecal injection of morphine 200 μg
  Other Names: M200
  Arms: Group II

SUMMARY:
Pruritus is the commonest side effect of intrathecal morphine especially in parturient, but the exact mechanism of pruritus is not clear. Many mechanisms have been suggested. Among these mechanisms is the activation of the 5-HT3 receptors by the intrathecally injected morphine.

DETAILED DESCRIPTION:
Forty parturients underwent elective cesarean section under spinal anesthesia were divided into two groups of 20 each in this prospective randomized study. Group I received 100 µg of intrathecal morphine (ITM) mixed with 12 mg of 0.5% heavy bupivacaine (M100) while group II received 200 µg of ITM mixed with 12 mg of 0.5% heavy bupivacaine (M200). Two blood samples were taken from each patient for serotonin estimation, preoperatively and 4 hrs later. Postoperatively all patients were assessed for pruritus (incidence & severity), visual analog scale (VAS), first request of analgesia, and total analgesic dose required within 24 hrs.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II term pregnant patients scheduled for elective cesarean section

Exclusion Criteria:

* patients with a known allergy to the study drugs
* significant cardiac, respiratory, renal, neurological, or hepatic disease; -coagulation disorders
* BMI > 30 kg/m2
* any itchy skin diseases.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2016-09-21 (Actual)

PRIMARY OUTCOMES:
Pruritus | 24 hours postoperative
  incidence
Pruritus | 24 hours postoperative
  severity

SECONDARY OUTCOMES:
serotonin | preoperative
  Serum level
serotonin | 4 hours postoperative
  Serum level

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed G Aly, M.D., Principal Investigator — Assiut university faculty of medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bonnet MP, Marret E, Josserand J, Mercier FJ. Effect of prophylactic 5-HT3 receptor antagonists on pruritus induced by neuraxial opioids: a quantitative systematic review. Br J Anaesth. 2008 Sep;101(3):311-9. doi: 10.1093/bja/aen202. Epub 2008 Jul 7. PMID 18611915